CLINICAL TRIAL: NCT01183182
Title: Confirmation of Clinical Effectiveness and Safety of CT-guided Percutaneous Lung Aspiration and Biopsy Performed With the Aid of the ActiSightTM Needle Guidance System
Brief Title: Safety and Effectiveness Study for a Needle Guidance System in Lung Biopsies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ActiViews Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: ACST-2010-1
Record Dates: First submitted 2010-08-13; First posted 2010-08-17 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2011-03

CONDITIONS: Lung Diseases
Keywords: Lung nodule; Lung lesion
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Needle Guidance (Experimental): Lung biopsies performed with the needle guidance system.
  Interventions: Device: ActiSight Needle Guidance System

INTERVENTIONS:
Device: ActiSight Needle Guidance System — Three different groups of patients defined per lesion size
  Other Names: CT-Guide Needle Guidance System

SUMMARY:
This study is designed to provide clinical data regarding safety and clinical effectiveness of the ActiSight Needle Guidance System in assisting radiologically guided percutaneous needle biopsy or aspiration of pulmonary lesions, which is a common procedure.

DETAILED DESCRIPTION:
This will be a prospective, single-arm study. At least three centers in Canada will participate in the study and at least 4 different experienced staff radiologists will perform the procedures for the study.

A total of forty eight (48) consecutive subjects meeting the eligibility criteria, scheduled for clinically indicated CT guided lung biopsy or aspiration procedure at the participating centers will be invited to enroll in the study. To ensure diversity in the study population, consecutive patients will be enrolled in the following groups until these groups are fully enrolled:

Lesion size ≥1.0 cm and ≤ 1.5 cm: 10 patients; Lesion size >1.5 and ≤ 3.0 cm: 19 patients; Lesion size >3.0 cm: 19 patients.

A maximum of 24 patients will be enrolled at each center.

Informed consent will be signed prior to the procedure. Subject data collection on the day of the procedure will include demographics, relevant medical history and vital signs. Enrolled subjects will undergo CT guided percutaneous lung aspiration and/or biopsy as clinically indicated by a qualified physician, utilizing the ActiSight Needle Guidance System. Subjects will be followed-up as outlined below to assess adverse events related to the procedure. A subject's enrollment in the study will be completed after the follow-up visit or after resolution of any procedure related adverse event.

A procedure difficulty classification is defined for this study, based on existing literature. Difficulty levels for all procedures will be recorded and included in the final report.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older at the time of enrollment;
* Subjects scheduled for clinically indicated CT guided percutaneous lung aspiration/biopsy;
* Written informed consent to participate in the study;
* Ability to comply with the requirements of the study procedures;
* Verified home address and phone number to facilitate study follow-up.

Exclusion Criteria:

* Significant coagulopathy that cannot be adequately corrected;
* Subjects who participated in an active stage of any drug, intervention or treatment trial within 30 days of enrollment;
* Subjects with preexisting conditions which, in the opinion of the investigator, interfere with the conduct of the study;
* Subjects who are uncooperative or cannot follow instructions;
* Mental impairment that may preclude completion of the study procedure;
* Pregnant or nursing female subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with successful targeting accuracy as defined by the frequency of placing the needle at a location suitable for obtaining tissue sample from the target lesion. | 30 to 60 minutes after starting the biopsy procedure
  Needle location suitable for obtaining tissue sample will be determined by a physician reviewing the CT images.
  All 48 subjects undergoing aspiration or biopsy procedures with the CT met the primary efficacy endpoint of placement of the procedure needle at a location suitable for obtaining a tissue sample from the target lesion as determined by the investigator (100%; 95% CI, 93-100%).

SECONDARY OUTCOMES:
Total CT-Guided procedure time Patient radiation exposure during the procedure Number of CT scans during the procedure | 30 to 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Paul Narinder, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - McGill University Health Center, Royal Victoria Hospital, Montreal General Hospital, Montreal, Quebec